CLINICAL TRIAL: NCT00878124
Title: The Influence of Concomitant Co Enzyme Q10 Use on Pregnancy Outcome in Intrauterine Insemination
Brief Title: How Dose Coenzyme Q10 Supplementation During Infertility Treatment Effects Pregnancy Outcome
Acronym: CoQ10
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Very low recruitment rate
Sponsor: University of Toronto (Other)
Collaborators: Toronto Centre for Advanced Reproductive Technology (Other); Ferring Pharmaceuticals (Industry)
Responsible Party: Dr. Yaakov Bentov, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CoQ10 - 08-0205-A
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Poor Ovarian Response
Keywords: Poor ovarian response; Chromosomal aberrations; poor pregnancy outcome; Late maternal age
MeSH Terms: conditions — Chromosome Aberrations | interventions — Ubiquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- CoQ10 (Experimental): Coenzyme Q10 co-treatment
  Interventions: Dietary Supplement: Coenzyme Q10 co treatment
- Placebo control (Placebo Comparator): Placebo Co-treatment
  Interventions: Other: Placebo Caps

INTERVENTIONS:
Dietary Supplement: Coenzyme Q10 co treatment — CoenzymeQ10 300mg twice a day continuously. Ceased when patient conceives or at the end of the study.
  Other Names: Ubiquinone.
  Arms: CoQ10
Other: Placebo Caps — 3 caps twice a day continuously until pregnant or at the end of the study.
  Arms: Placebo control

SUMMARY:
As women age the ovarian response and pregnancy rate are reduced while the rate of chromosomal abnormalities in the embryos is increased. Oocyte maturation, accurate chromosomal segregation as well as early embryo development and implantation are dependent on the supply of large amounts of energy, which unlike other cells can only arise from the mitochondria. With age the mitochondria becomes less efficient due to damage to its unique DNA, resulting in decreased energy production. The proposed study will examine the effect of the combination of a dietary supplement, Co enzyme Q10 on pregnancy rate and response of the ovaries to a medication that stimulates follicle growth. The investigators hypothesize that the improved energetic state of the oocyte would result in a more accurate chromosomal separation, increased embryo quality and pregnancy rate.

DETAILED DESCRIPTION:
The study will be organized on an outpatient basis at the Toronto Centre for Advanced Reproductive Technology (TCART) and at the Lifequest Centre for Reproductive Medicine. The study will involve 100 women aged 38-43 years.

In the first cycle, study participants will be randomly assigned to either placebo or COQ10 capsules, (AOR - Advanced Orthomolecular Research Inc. 19 St NE Calgary, Alberta, NHPD registration codes 135307 and 113519, respectively). Study participants will take 600 mg of CoQ10 orally or identical placebo capsules for up to 5 cycles if pregnancy does not occur. All subjects will commence controlled ovarian stimulation (COH) using highly purified human menopausal gonadotropins (Menopur; Ferring Inc., North York,Ontario Canada). The starting dosage of Menopur will range from 75IU to 250 IU daily S.C. will be determined by the physician and will begin on the third day of menses, and will continue until the day prior to human chorionic gonadotropin (hCG) administration. The dosage will not be changed and must be maintained for the duration of the study. Menopur will continue daily until follicular development is considered adequate. (at least 1 follicle is >17 mm, and the E2 level is acceptable for the number of follicles present). The patient will receive an injection of hCG 250 mcg (Ovidrel, EMD Serono,Oakville, Ontario, Canada ), SC for the final stage of follicular maturation. Insemination will be by intrauterine insemination (IUI). Luteal support will consist of progesterone suppositiories 200mg (Kingsway Pharmacy,Toronto, Ontario Canada) vaginally per day starting on the day of IUI and will continue for 2 weeks until the serum beta hCG result. At the end of each cycle serum beta hCG will be drawn and if women are pregnant CoQ10/ placebo will be discontinued. If pregnant, luteal support will continue until 10 weeks gestation. If the patient is not pregnant she will have a cycle off COH but may attempt to conceive naturally. In the third cycle, COH using the same dose of Menopur as in the first cycle will be performed with IUI as in cycle one. If not pregnant, another cycle off treatment will be followed by the fifth cycle in which COH and IUI is performed..

The study endpoints will be:

1. Primary outcome measure will be pregnancy rate.
2. Secondary outcome measures will include:

   * Peak estradiol level
   * The number of follicles > 14 mm on day of hCG
   * Number of days of stimulation / units of Menopur needed

ELIGIBILITY:
Inclusion Criteria:

* Each patient must meet the following criteria:
* Age 38-43 years at the time of enrollment
* Diagnosis of primary infertility

Exclusion Criteria:

* Patients must NOT have any of the following:
* Body mass index (BMI) > 38 kg/m2
* Early follicular phase (day 2-4) serum FSH level > 20 mIU/ml.
* Abnormal uterine cavity and /or tubal blockage as evidenced by sonohysterogram or hysterosalpingography
* Any current use of systemic steroid medication within 3 months of study enrollment.
* Any contraindication to being pregnant and carrying a pregnancy to term.
* Contraindication for the use of CoQ10, Menopur, hCG, and Prometrium.
* Any ovarian or abdominal abnormality that may interfere with adequate TVS evaluation.
* Absence of one ovary
* Clinically relevant systemic disease (e.g., Insulin-dependent diabetes, adrenal dysfunction, organic intracranial lesion, hyperprolactinemia, or hypothalamic tumor) or serious illness (Neoplasia).
* History (within past 12 months) or current abuse of alcohol or drugs.
* Administration of any investigational drugs within three months prior to study enrollment.
* Any medical condition that may interfere with the absorption, distribution, metabolism or excretion of the study drugs, gastrointestinal diseases, mal absorption syndromes and liver dysfunction
* Unexplained gynecological bleeding.
* Abnormal sperm quality or semen sample inadequate for IUI preparation (TMC > 1x106 post wash)
* Patient not able to communicate adequately with the investigators and to comply with the requirements of the entire study.
* Abnormal COH screening bloods for either partner, including: HIV serology, Hepatitis B and C serology, Rubella, and syphilis serology prior to participation in study.
* Unwillingness to give written informed consent.
* The concurrent use of any of the following drugs:
* CoQ10: Daunorubicin, Doxorubicin, Blood Pressure Medications, Warfarin, Timolol, atorvastatin, cerivastatin, lovastatin, pravastatin, simvastatin gemfibrozil, tricyclic antidepressant medications (including amitriptyline, amoxapine, clomipramine, desipramine, doxepin, imipramine, nortriptyline, protriptyline, and trimipramine).

Ages: 38 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-06

PRIMARY OUTCOMES:
Pregnancy rate | Every cycle

SECONDARY OUTCOMES:
Peak estradiol level | Every cycle
The number of follicles > 14 mm on day of hCG | Every cycle
Number of days of stimulation/units of Menopur needed | Every cycle

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Casper, Prof, Principal Investigator — University of Toronto
Locations (2):
- Canada (2):
  - LifeQuest Centre for Reproductive Medicine, Toronto, Ontario
  - Toronto center for advanced reprodutive technology, Toronto, Ontario